CLINICAL TRIAL: NCT01138501
Title: A Multi-Centre, Open-Label, Non-Controlled Trial on Safety and Efficacy of N8 in Previously Treated Paediatric Patients With Haemophilia A
Brief Title: Safety and Efficacy of Turoctocog Alfa in Previously Treated Male Children With Haemophilia A
Acronym: guardian™ 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7008-3545; U1111-1113-7182 (Other: WHO); 2009-016383-36 (EudraCT Number); NCT01250028 (obsolete NCT alias)
Record Dates: First submitted 2010-05-28; First posted 2010-06-07 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-02

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII N8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rFVIII (Experimental)
  Interventions: Drug: turoctocog alfa

INTERVENTIONS:
Drug: turoctocog alfa — Subjects will be treated 3 times per week or every second day with intravenous injections of turoctocog alfa. The dose range for preventive treatment is 25-60 IU/kg body weight depending on treatment regimen.
Drug: turoctocog alfa — Subjects will undergo half-life evaluation of their current factor VIII product and pharmacokinetic session with turoctocog alfa before entering preventive treatment (subjects with available evaluation of terminal half-life within the last year are to be excluded from receiving factor VIII). Intravenous injections. The dose range for preventive treatment is 25-60 IU/kg body weight depending on treatment regimen.

SUMMARY:
This trial is conducted in Asia, Europe, and North and South America. The aim of this clinical trial is to investigate the safety and efficacy of turoctocog alfa (recombinant factor VIII, rFVIII (N8)) in male previously treated paediatric subjects with haemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with severe (baseline FVIII less than or equal to 1%) haemophilia A
* Age below 12 years and weight at least 11 kg

Exclusion Criteria:

* Surgery planned to occur during trial participation (exceptions are port placement, dental extractions, and minor, uncomplicated emergent procedures)
* Congenital or acquired coagulation disorders other than haemophilia A
* Any history of FVIII inhibitors (greater than or equal to 0.6 BU/mL)

Max Age: 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (38):
- United States (18):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Torrance, California
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Augusta, Georgia
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, East Lansing, Michigan
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Brooklyn, New York
  - Novo Nordisk Investigational Site, Valhalla, New York
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
- Brazil (4):
  - Novo Nordisk Investigational Site, Curitiba, Paraná
  - Novo Nordisk Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Novo Nordisk Investigational Site, Campinas, São Paulo
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
- Novo Nordisk Investigational Site, Milan, Italy
- Novo Nordisk Investigational Site, Shizuoka-shi, Shizuoka, Japan
- Novo Nordisk Investigational Site, Vilnius, Lithuania
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Poland (2):
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- Novo Nordisk Investigational Site, San Juan, Puerto Rico
- Russia (2):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
- Novo Nordisk Investigational Site, Belgrade, Serbia
- Novo Nordisk Investigational Site, Taipei, Taiwan
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Bornova-IZMIR
  - Novo Nordisk Investigational Site, İzmit

REFERENCES:
- [Result] Kulkarni R, Karim FA, Glamocanin S, Janic D, Vdovin V, Ozelo M, Rageliene L, Carboni E, Laguna P, Dobaczewski G, Seremetis S, Lindblom A, Santagostino E. Results from a large multinational clinical trial (guardian3) using prophylactic treatment with turoctocog alfa in paediatric patients with severe haemophilia A: safety, efficacy and pharmacokinetics. Haemophilia. 2013 Sep;19(5):698-705. doi: 10.1111/hae.12165. Epub 2013 May 8. PMID 23651313
- [Result] Santagostino E, Lentz SR, Misgav M, Brand B, Chowdary P, Savic A, Kilinc Y, Amit Y, Amendola A, Solimeno LP, Saugstrup T, Matytsina I. Safety and efficacy of turoctocog alfa (NovoEight(R)) during surgery in patients with haemophilia A: results from the multinational guardian clinical trials. Haemophilia. 2015 Jan;21(1):34-40. doi: 10.1111/hae.12518. Epub 2014 Oct 2. PMID 25273984
- [Result] Ozelo MC. Updates from guardian: a comprehensive registration programme. Eur J Haematol. 2015 Dec;95 Suppl 81:22-9. doi: 10.1111/ejh.12648. PMID 26679394
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of a total of 39 initiated trial sites, 26 sites enrolled and dosed at least one patient. The country distribution was as follows: Brazil (3), Italy (1), Lithuania (1), Macedonia (1), Malaysia (1), Poland (2), Russia (2), Serbia (1), Taiwan (1), Turkey (3) and the United States of America (10).
Groups:
- All Subjects Treated With Turoctocog Alfa: The patients received bleeding preventive treatment with a single dose of turoctocog alfa of 25-50 IU/kg every second day or 25-60 IU/kg three times weekly. Turoctocog alfa was administered as a slow bolus i.v. injection (approximately 1-2 mL/min). Pharmacokinetic assessments were performed in at least 13 patients from each age cohort. Each patient participating in the pharmacokinetic assessments received one dose of previous factor VIII (FVIII) and one dose of turoctocog alfa.
Period: Overall Study
Arm/Group | All Subjects Treated With Turoctocog Alfa
Started | 65 (Two subjects withdrew consent after being enrolled but before receiving any trial product.)
Exposed | 63
Completed | 60
Not Completed | 5
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects Treated With Turoctocog Alfa
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.08 (2.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 63
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 47
Region of Enrollment [Number; unit: participants]
  Brazil | 9
  Serbia | 5
  Italy | 2
  Lithuania | 4
  Macedonia, The Former Yugoslav Republic of | 5
  Malaysia | 5
  Poland | 5
  Russia | 8
  Taiwan | 1
  Turkey | 7
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: The Incidence Rate of FVIII Inhibitors (Greater Than or Equal to 0.6 Bethesda Units (BU))
Description: The incidence rate of FVIII inhibitors was calculated by including all patients with inhibitors in the nominator and including all patients with a minimum 50 exposure plus any patients with less than 50 exposures but with inhibitors in denominator.
Time Frame: The adverse events were collected throughout the trial, corresponding to an average of 138 days per subject.
Population: The safety analysis set includes all 63 subjects who received at least one dose of the investigational product. The analysis of the primary endpoint included all subjects with at least 50 exposure days and/or with inhibitors. A total of 59 subjects had 50 exposure days (EDs).
Measure: Number; unit: N with Inhibitors / N with ≥50 EDs
Arm/Group | All Subjects Treated With Turoctocog Alfa
Number analyzed (Participants) | 59
N with Inhibitors / N with ≥50 EDs | 0

2. Secondary Outcome: Frequency of Adverse Events (AEs)
Description: Adverse event was defined as events occurring after administration of trial product. Severe AEs: considerable interference with subject's daily activities, unacceptable. Moderate AEs: Marked symptoms, moderate interference with the patient's daily activities. Mild AEs: No or transient symptoms, no interference with the patient's daily activities. Serious AE: AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: The adverse events were collected throughout the trial, corresponding to an average of 138 days per subject
Population: Safety analysis set includes all subjects who received at least one dose of the investigational product.
Measure: Number; unit: events
Arm/Group | All Subjects Treated With Turoctocog Alfa
Number analyzed (Participants) | 63
events
  All AEs | 86
  Severe AEs | 0
  Moderate AEs | 11
  Mild AEs | 74
  Serious AEs | 3
  Probably or possibly related | 2

ADVERSE EVENTS:
Time Frame: The adverse events were collected throughout the trial, corresponding to an average of 138 days per subject.
Description: Safety analysis set includes all subjects who received at least one dose of the investigational product.
Arm/Group | All Subjects Treated With Turoctocog Alfa
Serious Adverse Events (participants affected / at risk) | 3/63
Other Adverse Events (participants affected / at risk) | 14/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects Treated With Turoctocog Alfa (N=63)
Device related infection (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects Treated With Turoctocog Alfa (N=63)
Vomiting (Gastrointestinal disorders) | 4 (4)
Nasopharyngitis (Infections and infestations) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 4 (4)
Headache (Nervous system disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol.